CLINICAL TRIAL: NCT01770964
Title: Evaluation of the Impact of Subject and Staff Training on the Pregabalin vs. Placebo Difference in Subjects With Painful Diabetic Neuropathy (PDN)
Brief Title: Evaluation of the Impact of Training on Outcome Measures in Subjects With Painful Diabetic Neuropathy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Analgesic Solutions (Industry)
Collaborators: Astellas Pharma Europe B.V. (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ALPMF-0007-2012
Record Dates: First submitted 2012-12-13; First posted 2013-01-18 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Diabetes Mellitus; Painful Distal Symmetric Sensorimotor Polyneuropathy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Training Type A, pregabalin (Other): Subjects randomized to receive pregabalin at a site that received training Type A
  Interventions: Drug: Pregabalin; Behavioral: Training Type A
- Training Type B, pregabalin (Other): Subjects randomized to receive pregabalin at a site that received training Type B
  Interventions: Drug: Pregabalin; Behavioral: Training Type B
- Training Type A, placebo (Other): Subjects randomized to receive placebo at a site that received training Type A
  Interventions: Drug: placebo; Behavioral: Training Type A
- Training Type B, placebo (Other): Subjects randomized to receive placebo at a site that received training Type B
  Interventions: Drug: placebo; Behavioral: Training Type B

INTERVENTIONS:
Drug: Pregabalin
  Arms: Training Type A, pregabalin; Training Type B, pregabalin
Drug: placebo
  Arms: Training Type A, placebo; Training Type B, placebo
Behavioral: Training Type A
  Arms: Training Type A, placebo; Training Type A, pregabalin
Behavioral: Training Type B
  Arms: Training Type B, placebo; Training Type B, pregabalin

SUMMARY:
The difference between active treatment and placebo in a clinical trial of an analgesic appears to depend on a variety of factors other than the actual efficacy of the drug itself, including various aspects of study design and conduct. One potential such factor is how information about the study is presented to research staff and patients. The purpose of this study is to examine the impact of different presentations of information on the difference between pregabalin and placebo observed in a clinical trial in patients with painful diabetic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Willingly signs and dates an Informed Consent Form (ICF) that is approved by an Institutional Review Board/Independent Ethics Committee (IRB/IEC), prior to the conduct of any study-specific procedures;
* Is at least 18 years old;
* Has a diagnosis of type 1 or type 2 diabetes and painful distal symmetric sensorimotor polyneuropathy;
* Has experienced a minimum duration of PDN of at least 6 months;
* Is on stable diabetic medication that is not expected to change during the study;
* Has a worst pain intensity over the past 24 hours as a 4 or higher on a 0-10 numerical rating scale at Screening;
* And is able to read and communicate meaningfully in English and comply with all study procedures

Exclusion Criteria:

* Has a psychiatric or psychological disorder that in the judgment of the Investigator would interfere with the completion of the study, confound the study results, or pose subject risk;
* Has an uncontrolled, clinically significant medical condition that in the judgment of the Investigator may contraindicate use of pregabalin or participation in the study (e.g., hepatic, respiratory, or hematologic illness; cardiovascular disease; or symptomatic peripheral vascular disease);
* Has experience as an investigator or a study staff member in clinical trials research in a role that involved direct patient contact;
* Participated in any of the following studies: Analgesic Solutions Protocol # ALPMF.SOW.0007, Analgesic Solutions Protocol # ALPMF.SOW.0007.02, or Astellas Protocol # E05-CL-3004;
* Has pain of other origin that might confound assessment of PDN;
* Has major skin ulceration;
* Has had an amputation other than toes;
* Has a history of suicide attempt within the past 1 year;
* Reports current suicidal ideation within the past 1month;
* Has history of kidney disease that is likely to decrease creatinine clearance;
* Has creatinine clearance below 60 as calculated by Cockroft-Gault equation for serum creatinine;
* Has a history of drug or alcohol abuse within the past 1 year;
* Has hypersensitivity, intolerance, or allergy to pregabalin or gabapentin;
* Subject is pregnant, is considering becoming pregnant during the study, is breastfeeding or unwilling to use adequate birth control during the study;
* Participated in another clinical trial within the past month;
* Is involved in an ongoing or settled worker's compensation claim, disability, or litigation;
* Has a known failure to respond to pregabalin or gabapentin at a clinically relevant dose due to either efficacy or tolerability;
* Or has taken opioids on an as-needed basis within 1week of Screening, or has taken pregabalin or gabapentin within 30 days of screening. Subjects on stable doses opioids, antidepressants, non-steroidal anti-inflammatory drugs, or low-dose aspirin will be allowed to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
change in pain severity rating | Screening/Visit 1 (Day 1) and Visit 4 (Day 15-18)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremiah J Trudeau, PhD, Principal Investigator — Analgesic Solutions
Locations (6):
- United States (6):
  - St. Elizabeth's Medica Center, Brighton, Massachusetts
  - MedVadis Research Corporation, Watertown, Massachusetts
  - Neuro Care Medical Associates, Johnson City, New York
  - University of Rochester, Rochester, New York
  - Blair Medical Associates, Inc., Altoona, Pennsylvania
  - Clinical Partners, Johnston, Rhode Island